CLINICAL TRIAL: NCT07406724
Title: Randomized, Controlled, Open-label Phase 2 Clinical Trial of HS-IT101 Injection Versus Chemotherapy for Patients With Advanced Melanoma
Brief Title: HS-IT101 Injection Versus Chemotherapy in the Treatment of Advanced Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qingdao Sino-Cell Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-IT101ST01-Ⅱ
Record Dates: First submitted 2026-02-02; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Melanoma (Excluding Uveal Melanoma)
Keywords: Advanced Melanoma
MeSH Terms: conditions — Melanoma | interventions — Toll-Like Receptor 1; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-IT101 monotherapy (Experimental): Tumor Tissue Sampling、Bridging Therapy、Lymphodepletion Conditioning、Infusion of HS-IT101 Injection、IL-2 Administration for Tumor-Infiltrating Lymphocyte (TIL) Therapy
  Interventions: Procedure: Tumor Tissue Sampling; Drug: Lymphodepletion Conditioning; Drug: Infusion of HS-IT101 Injection; Drug: IL-2 Administration for Tumor-Infiltrating Lymphocyte (TIL) Therapy
- Investigator's Choice of Chemotherapy Regimens (Active Comparator)
  Interventions: Drug: Investigator's selection of appropriate chemotherapy regimen

INTERVENTIONS:
Procedure: Tumor Tissue Sampling — Surgical procurement of the subject's tumor tissue for autologous tumor-infiltrating lymphocyte (TIL) preparation
  Arms: HS-IT101 monotherapy
Drug: Lymphodepletion Conditioning — Intravenous Infusion of Cyclophosphamide and Fludarabine
  Arms: HS-IT101 monotherapy
Drug: Infusion of HS-IT101 Injection — Single intravenous infusion of HS-IT101 Injection following lymphodepletion conditioning
  Arms: HS-IT101 monotherapy
Drug: IL-2 Administration for Tumor-Infiltrating Lymphocyte (TIL) Therapy — Subcutaneous injection of IL-2 following intravenous infusion of HS-IT101 Injection
  Arms: HS-IT101 monotherapy
Drug: Investigator's selection of appropriate chemotherapy regimen — Single-agent or combination chemotherapy regimens include dacarbazine, temozolomide, paclitaxel, and carboplatin.
  Arms: Investigator's Choice of Chemotherapy Regimens

SUMMARY:
This is a multicenter, randomized controlled, open-label Phase II clinical study designed to evaluate the efficacy and safety of HS-IT101 Injection versus the investigator's choice of chemotherapy in participants with advanced melanoma. A total of 90 participants are planned to be enrolled, and eligible participants will be randomly assigned to the experimental group or control group at a 1:1 ratio. The experimental group will receive a single administration of autologous tumor-infiltrating lymphocyte therapy, while the control group will receive chemotherapy regimens selected by the research physicians. Efficacy and safety evaluations will be conducted for all enrolled participants throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 75 years, inclusive.
2. Patients with cytologically or histologically confirmed unresectable advanced, recurrent, or metastatic melanoma (excluding uveal melanoma), who have experienced disease progression after failure of systemic therapy recommended in the 2025 CSCO Guidelines.
3. Disease Progression Following Anti-PD-1 Therapy.
4. At least one tumor lesion not treated with radiotherapy or other local therapies within 28 days prior to resection, suitable for autologous tumor-infiltrating lymphocyte (TIL) preparation, with a minimum tissue weight of ≥0.050 g.
5. At least one measurable tumor lesion per RECIST 1.1 after tumor tissue sampling.
6. ECOG performance status ≤ 1.
7. Expected survival ≥ 3 months.
8. Adequate organ and bone marrow function as confirmed by screening assessments.
9. Documented by echocardiography showing left ventricular ejection fraction (LVEF) ≥50%；Absence of arrhythmia requiring therapeutic intervention；Electrocardiogram (ECG) criteria；QT interval corrected by Frederica's formula (QTcF) ≤470 ms；Baseline peripheral oxygen saturation (SpO₂) >91% in room air.
10. Adverse reactions from prior therapy have resolved to CTCAE v5.0 grade ≤1 before randomization, except for hypothyroidism and alopecia judged by the investigator as non-safety concerns.
11. Effective non-pharmacological contraceptive measures must be used from the signing of the informed consent form until 1 year after TIL cell infusion.
12. The subject fully understands the trial, voluntarily provides written informed consent, and is able to comply with scheduled visits and protocol-specified procedures.

Exclusion Criteria:

1. Patients with a history of severe hypersensitivity reactions (e.g., anaphylaxis, Stevens-Johnson syndrome, or toxic epidermal necrolysis) to any component of the following agents.
2. Presence of any uncontrolled clinical conditions, including but not limited to:

   * Poorly controlled hypertension (systolic BP ≥160 mmHg and/or diastolic BP ≥100 mmHg at rest despite antihypertensive therapy);
   * Congestive heart failure (NYHA Class III/IV).
3. History of deep vein thrombosis (DVT) or pulmonary embolism (PE); myocardial infarction; severe or unstable arrhythmia or angina; percutaneous coronary intervention, acute coronary syndrome, or coronary artery bypass grafting; cerebrovascular accident, transient ischemic attack, or cerebral embolism within the past 6 months.
4. Active autoimmune diseases requiring systemic therapy during the study period（Subjects with the following conditions may be enrolled：Eczema, vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic therapy within the last 2 years and not expected to recur, or other autoimmune diseases under stable control;Hypothyroidism requiring only thyroid hormone replacement;Type 1 diabetes requiring only insulin replacement therapy.）
5. Organ transplant or history of hematopoietic stem cell transplantation.
6. Use of systemic immunosuppressive agents (e.g., corticosteroids) within 4 weeks prior to randomization, or presence of comorbid conditions requiring such medications during the trial period.Exception: Intranasal or topical corticosteroids are permitted.
7. Receipt of systemic anti-tumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to randomization, or planned participation in another interventional clinical trial during the study period.
8. Acute or chronic infections, including:

   * HIV-positive status, Treponema pallidum antibody positivity, or clinically active hepatitis B or C(Note: For hepatitis B, HBsAg- or HBeAg-positive individuals with HBV DNA below the lower limit of normal at the study site may be enrolled; for hepatitis C, HCVAb-positive individuals with HCV RNA below the lower limit of normal at the study site may be enrolled);
   * Active infections requiring systemic therapy or active tuberculosis infection.
9. Subjects who received any live attenuated vaccine within 3 months prior to screening or planning to receive live vaccines during the trial period.
10. Subjects who have undergone major organ surgery or experienced clinically significant trauma within 4 weeks prior to screening, or require elective surgery during the trial period.
11. Patients presenting with pre-screening surgical complications or delayed wound healing, and deemed by the investigator to confer increased risks during lymphodepleting pretreatment, adoptive TIL therapy, and high-dose IL-2 adjuvant therapy.
12. Patients with a history of other primary malignancies diagnosed within 5 years prior to screening are excluded, except for radically treated basal cell carcinoma, squamous cell carcinoma of the skin, and/or carcinoma in situ.
13. Patients with severe respiratory diseases (including but not limited to a documented history of or concurrent severe interstitial lung disease (ILD), severe chronic obstructive pulmonary disease (COPD), profound pulmonary insufficiency, or symptomatic bronchospasm).
14. Patients requiring surgical intervention for gastrointestinal hemorrhage, localized intestinal ischemia, or intestinal perforation.
15. Patients with symptomatic central nervous system (CNS) metastases
16. Patients with clinical symptoms of central nervous system (CNS) metastases who have received prior therapy for brain metastases and maintained radiographic stability (confirmed by MRI) for at least 12 weeks may be enrolled.
17. Pregnant or lactating women.
18. Individuals with a known history of psychiatric disorders, alcoholism, drug abuse, or substance abuse, as well as any other conditions deemed unsuitable for participation by the investigator .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 1 year
  Progression-Free Survival (PFS) assessed by Independent Review Committee (IRC)

SECONDARY OUTCOMES:
OS | 1 year
  Time from randomization to death from any cause, as well as 6-month and 12-month Overall Survival (OS) rates
ORR | 1 year
  Proportion of subjects with best overall response (BOR) of either partial response (PR) or complete response (CR)
DCR | 1 year
  Proportion of subjects with best response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) among total evaluable cases
DOR | 1 year
  The time from first documentation of complete response (CR) or partial response (PR) to first documented progressive disease (PD) or all-cause death, whichever occurs first
TTR | 1 year
  Time to First Response (TTR) from randomization in participants with a best overall response (BOR) of Complete Response (CR) or Partial Response (PR)
PFS | 1 year
  Progression-Free Survival (PFS) assessed by Investigator

IPD SHARING:
Plan to Share IPD: No